CLINICAL TRIAL: NCT06808685
Title: Real-world Multicenter National Study to Evaluate the Effectiveness and Safety of Biosimilar Bevacizumab Elovie in First-line Treatment in Participants With Unresectable Metastatic Colorectal Cancer
Brief Title: Real World Multicenter National Study to Evaluate the Effectiveness and Safety of Biosimilar Bevacizumab Elovie
Status: Recruiting | Type: Observational
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Other Study IDs: LB2401
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Elovie; bevacizumab; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer is one of the most common tumors and is the second most prevalent cause of cancer death, leading to almost 1 million deaths per year.Elovie is a bevacizumab biosimilar medicine marketed by Libbs Farmacêutica, which had its registration approved by ANVISA in May 2022.At the time of registration a robust evidence package was presented that included, for example, pharmacokinetic bioequivalence studies in patients with metastatic RCC (mRCC) and a phase III study in participants with non-small cell lung cancer .Conducting a real-world study to evaluate the effectiveness and safety of bevacizumab biosimilar Elovie in patients with mCRC is crucial to provide relevant information on how this therapy behaves in real-world clinical conditions in brazilian population.

DETAILED DESCRIPTION:
Observational, multicenter study with real-world data from specialized cancer centers in Brazil. Participants over 18 years of age, of both sexes, with unresectable clinical stage IV metastatic colorectal cancer, who have received Elovie® (bevacizumab biosimilar) at participating centers and who meet the eligibility criteria will be invited to participate. In this study, data on the effectiveness and safety of treatment with Elovie, as well as clinical and demographic characteristics and treatment patterns will be collected.

Participants will undergo standard treatment and clinical follow-up as determined by the treating physician.

Data collection will be performed by the researcher and the data transcribed into the Case Report Form data collection form designed specifically for the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes aged 18 years or older at the start of treatment with bevacizumab;
* Participants diagnosed with metastatic colorectal cancer, clinical stage IV, unresectable, by clinical definition in medical records, according to the investigator's assessment at the initial consultation and before any type of palliative treatment;
* Participants who are undergoing first-line treatment with Elovie and who have completed at least 1 cycle of treatment or participants who have started first-line treatment with another bevacizumab (reference or another biosimilar other than Elovie) but who have currently switched to Elovie and completed at least 1 cycle of treatment with it, and whose data is available at the institution participating in the study;
* Participants with the capacity to understand and consent to their participation in the study through the Free and Informed Consent Form

Exclusion Criteria:

* Participants who use or have used bevacizumab in a manner different from that described in the current version of the Elovie® package insert;
* Participants who have been treated with Elovie for a period longer than 12 treatment cycles;
* Participants who have started first-line treatment with another bevacizumab (reference or another biosimilar other than Elovie) and have completed more than 2 treatment cycles with it;
* Participants with a concomitant diagnosis of another active malignant neoplasm other than metastatic colorectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants of both sexes diagnosed with metastatic colorectal cancer, clinical stage IV unresectable, by clinical definition in medical records, according to the investigator's assessment at the initial consultation and before any type of palliative treatment.
Sampling Method: Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of treatment with bevacizumab | 24 months
  Median duration in months and number of cycles of first-line treatment until the switch to second-line treatment, for any reason, through the collection of electronic medical record data.

SECONDARY OUTCOMES:
progression-free survival | 24 months
  progression-free survival will be defined as the median time (in months) from the first dose of bevacizumab to disease progression
Overall survival | 24 months
  Overall survival will be defined as the median time (in months) from the first dose of bevacizumab until the occurrence of death, from any cause, during the 24-month follow-up period
The survival rate | 24 months
  The survival rate will be defined as the number and proportion of participants who remained alive after 24 months of follow-up
Objective Response Rate | 24 months
  The Objective Response Rate will be defined as the number and percentage of participants who had a Complete Response or Partial Response, using the usual methodology of the research center, during 24 months of follow-up after the start of bevacizumab use. The number and percentage of participants who had Stable Disease or Disease Progression will also be evaluated.
Functional capacity | 24 months
  Functional capacity will be assessed using the ECOG (Eastern cooperative oncology group) scale during 24 months of follow-up after starting bevacizumab.
  Scale ECOG Grade 0 - Fully active, able to carry on all pre disease performance without restriction Grade 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work Grade 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours Grade 3 - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours Grade 4 - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair Grade 5 - Dead https://ecog-acrin.org/resources/ecog-performance-status/
Safety assessment | 24 months
  To assess the occurrence of adverse events in the 24-month follow-up period since the first dose of Elovie.Assess the median duration of treatment through time in months and number of cycles until switching to another treatment other than the first line, for reasons of toxicity (adverse event).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Dor de Pesquisa E Ensino, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided